CLINICAL TRIAL: NCT05746832
Title: Failed Retrograde Cholangiopancreatography (ERCP) Stone Extraction: Surgical Interference Versus Follow up on Stent.
Brief Title: Failed Retrograde Cholangiopancreatography (ERCP) Stone Extraction: Surgical Interference
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zyad Osama Harith, Zyad Osama Harith Abulatif (General surgery resident), Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBD stones managment by ERCP
Record Dates: First submitted 2021-11-01; First posted 2023-02-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Common Bile Duct Calculi
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One session application of (ERCP) in the management of common bile duct stones. (Active Comparator): One session application of endoscopic stenting retrograde cholangiopancreatography (ERCP) in the management and clearance of difficult common bile duct stones and assessment of the differences in stone size and the largest CBD diameter before and after stenting in one or two sessions. Stone clearance and complications were also determined with the ERCP, and factors associated with complete clearance were evaluated in patients with difficult CBD stones (a large [≥ 20 mm] or multiple [≥ 3 sized ≥ 15 mm] CBD stones). And also compared the outcomes with conventional procedure of open surgery.
  Interventions: Procedure: Endoscopic stenting Retrograde Cholangiopancreatography (ERCP)
- Two sessions application of (ERCP) in the management of common bile duct stones. (Active Comparator): Two sessions application of endoscopic stenting retrograde cholangiopancreatography (ERCP) in the management and clearance of difficult common bile duct stones.and assessment of the differences in stone size and the largest CBD diameter before and after stenting in one or two sessions. Stone clearance and complications were also determined with the ERCP, and factors associated with complete clearance were evaluated in patients with difficult CBD stones (a large [≥ 20 mm] or multiple [≥ 3 sized ≥ 15 mm] CBD stones). And also compared the outcomes with conventional procedure of open surgery.
  Interventions: Procedure: Endoscopic stenting Retrograde Cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic stenting Retrograde Cholangiopancreatography (ERCP) — Assessment of the differences in stone size and the largest CBD diameter before and after stenting in one or two sessions. Stone clearance and complications were also determined with the ERCP, and factors associated with complete clearance were evaluated in patients with difficult CBD stones (a large [≥ 20 mm] or multiple [≥ 3 sized ≥ 15 mm] CBD stones). And also compared the outcomes with conventional procedure of open surgery.

SUMMARY:
Assessment of the differences in stone size and the largest CBD diameter before and after stenting in one or two sessions. Stone clearance and complications were also determined with the ERCP, and factors associated with complete clearance were evaluated in patients with difficult CBD stones (a large [≥ 20 mm] or multiple [≥ 3 sized ≥ 15 mm] CBD stones). And also compared the outcomes with conventional procedure of open surgery.

DETAILED DESCRIPTION:
Gallstones are a very common problem in developed countries. Most patients with gallstones remain asymptomatic throughout their lifetime, but 10 % - 25 % of them may develop biliary pain or complications, with an annual risk of about 2 % - 3 % for symptomatic disease and 1 % - 2 % for major complications. The development of symptomatic disease and complications is mostly related to the migration of stones into the common bile duct (CBD). Common bile duct stones (CBDSs) may be treated by endoscopic retrograde cholangiopancreatography (ERCP) or surgically during cholecystectomy. Removal of common bile duct (CBD) stones can still be difficult in patients with large or multiple stones despite an adequate sphincterotomy. Procedures such as mechanical, extracorporeal, electrohydraulic or laser lithotripsy, and chemical dissolution have been introduced as effective therapeutic interventions for irretrievable CBD stones. However, these techniques have their drawbacks, are not widely available, or are still under clinical evaluation. Several studies have shown that insertion of an endoscopic biliary stent is a safe, effective, and widely available measure. An indwelling stent provides biliary drainage and fragments large stones, thereby reducing the risk of cholangitis and allowing stones to pass spontaneously or rendering them more extractable at a later procedure. Thus, this study intends to shed a light on advances in diagnosis and management in patients with biliary difficult stones.

ELIGIBILITY:
Inclusion Criteria:

1. All cases of difficult common bile duct stones leading to variable occlusion.
2. Patients fit for intervention.
3. Patients informed consent for study.

Exclusion Criteria:

1. Surgically unfit cases according to ASA
2. Locally advanced irresectable cases.
3. Patients refuse consent to participate in the study.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time of procedure. | On the day of determined procedure.
  This is measured in hours.
Rate of stone size reduction. | Baseline.
  This is measured in millimeters.
Width of CBD. | Baseline.
  This is measured in millimeters.
Degree of stone clearance and complications. | Baseline.
  Those are determined by close monitoring of patients whether after ERCP or surgery.
Postoperative morbidity and mortality. | Baseline.
  Those are measures in percentage of patients in the study.

SECONDARY OUTCOMES:
Blood loss during the procedure. | Baseline.
  This is measured in milliliters.
Postoperative wound infection. | Baseline.
  This is measured in percentage of patients in the study.
Postoperative hospital stay. | Baseline.
  This is measured in days.
Postoperative hemorrhage. | Baseline.
  This is measured in milliliters.
Postoperative 30 day mortality rate. | Baseline.
  This is measured in percentage of patients in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Ali Ryad, Prof., Principal Investigator — Assiut University
Locations (1):
- Assiut universty Hospital, Asyut, Egypt